CLINICAL TRIAL: NCT01798095
Title: A Randomized, Double-blind, Equivalence Study of the Specificity of Tuberculin Purified Protein Derivative (PPD) (Aplisol®) in Comparison With a Reference Standard
Brief Title: Equivalence Study of Specificity of PPD
Acronym: 03
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JHP Pharmaceuticals LLC (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: JHP-03
Record Dates: First submitted 2013-01-31; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Tuberculosis Infection
Keywords: TB, Aplisol
MeSH Terms: conditions — Latent Tuberculosis | interventions — Tuberculin; Reference Standards

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aplisol (Experimental): To confirm the response of PPD materials
  Interventions: Biological: Aplisol@ PPD material; Biological: Reference Standard
- PPD Standard (Active Comparator): Determine equivalent specificity for new material compared to standard material.
  Interventions: Biological: Aplisol@ PPD material; Biological: Reference Standard

INTERVENTIONS:
Biological: Aplisol@ PPD material — Determine equivalency of materials
  Other Names: Aplisol@
Biological: Reference Standard — Reference standard material for comparison to newly produced materials.
  Other Names: US Reference Standard

SUMMARY:
Determine if investigational products and reference standard produce similar responses.

DETAILED DESCRIPTION:
Primary:

To determine if the 2 investigational products (Aplisol formulated from the new Tuberculin PPD drug substance and the reference standard PPD-S2) produce qualitatively similar responses (positive or negative) in subjects who are uninfected with M. tuberculosis (Mtb) or other mycobacteria.

Secondary:

1. To determine if the 2 investigational products have equivalent specificity for detecting subjects currently or previously infected with Mtb;
2. To assess the tolerability of the investigational products in terms of the local and systemic reactogenicity events.

ELIGIBILITY:
Inclusion Criteria:

* Males or nonpregnant females, age 18 to 70 years

  * Negligible risk of manifesting a positive PPD test as evidenced by:

    * Prior history of negative PPD test or interferon gamma release assay (IGRA) within 14 months before Screening
    * No history of Bacillus Calmette- Guérin vaccination; or if vaccination status is uncertain, was born in the US and did not live outside the US as a child
    * No history of Mtb or Mtb therapy (including isoniazid, rifampin, ethambutol, pyrazinamide, or streptomycin)
    * No history of infection with atypical mycobacteria, including suspicious chest roentgenogram
    * No history of high risk medical conditions (eg, HIV infection or other immunosuppressive conditions, severe chronic renal disease [as evidenced by a creatinine clearance < 30 ml/min], poorly controlled diabetes mellitus, silicosis, intravenous drug use, or alcohol abuse)
    * No known close contact to a confirmed Mtb case (family or social setting)
    * No history of living or travelling in India, China, Sub-Saharan Africa, or Southeast Asia in the past 6 months
    * No exposure (other than casual) to high-risk environments for Mtb exposure (eg, prisons, homeless shelters); healthcare workers are allowed

Exclusion Criteria:

* Subject is of childbearing potential and unable to use contraceptives; is planning pregnancy; is pregnant or lactating

  * History of anaphylactic type reaction or other severe reaction to PPD in the past, including a history of blistering or sloughing
  * Presence of conditions that may suppress TST reactivity, including:

Protocol No. JHP-Aplisol-03 Confidential 04 May 2012 Page 8 of 38

* Acute viral infections, including measles, mumps, chicken pox, human immunodeficiency virus (HIV1, HIV2). Mild viral syndromes are allowed.
* Acute bacterial infections including typhoid fever, brucellosis, typhus, leprosy, or pertussis
* Acute systemic fungal infection
* Live virus vaccinations within the past 6 weeks, including measles, mumps, polio, varicella, or FluMist®
* Metabolic derangements (eg, poorly controlled diabetes, Cushing syndrome, chronic renal failure [as evidenced by a creatinine clearance < 30 ml/min])

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Determination of similarity in responses | 72 hours
  To determine if the 2 investigational products (Aplisol formulated from the new Tuberculin PPD drug substance and the reference standard PPD-S2) produce qualitatively similar responses (positive or negative) in subjects who are uninfected with M. tuberculosis (Mtb) or other mycobacteria.Skin test responses will be used to determine product similarity in responses.

SECONDARY OUTCOMES:
Determine equivalent specificity | 72 hours
  To determine if the 2 investigational products have equivalent specificity for detecting subjects currently or previously infected with Mtb; 2) To assess the tolerability of the investigational products in terms of the localand systemic reactogenicity events. Skin responses to new PPD and reference standard will be monitored to determine equivalent specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States